CLINICAL TRIAL: NCT01074151
Title: The Cymbalta Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Other Study IDs: 12938; F1J-MC-B034 (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy
Keywords: Pregnancy; pregnant; Cymbalta; Pregnancy Outcomes
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pregnant patients exposed to Cymbalta: Pregnant patients exposed to Cymbalta (duloxetine) at any time during pregnancy, beginning on or after the first day of the last menstrual period
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — any exposure to duloxetine that occurred during pregnancy

SUMMARY:
The Cymbalta Pregnancy Registry is a U.S. based Registry designed to monitor women who are exposed to Cymbalta (duloxetine) during pregnancy. This is an observational, exposure-registration and follow-up registry.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient evidence (e.g., date or gestational age) to confirm that Cymbalta exposure occurred during pregnancy
* Sufficient data to establish in which trimester of pregnancy the exposure to Cymbalta first occurred (i.e., first, second or third trimester)
* Sufficient information to determine whether the pregnancy is prospectively or retrospectively registered (i.e., whether the outcome of pregnancy was known at the time of first contact with the Registry)
* Date the pregnancy exposure is reported to the Registry
* Source of the report (Health Care Professional or pregnant patient)
* Full contact information for the reporter and Health Care Professional willing and able to provide accurate pregnancy-related information (name, address, phone number, etc.)

Exclusion Criteria:

* Reported cases that do not meet the minimum criteria for Registry enrollment are deemed ineligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant patients exposed to Cymbalta (duloxetine) at any time during pregnancy, beginning on or after the first day of the last menstrual period
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2009-07; Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
To estimate the risk of major congenital anomalies among pregnancies exposed to Cymbalta | maximum of 22 months

SECONDARY OUTCOMES:
To estimate risk of recognized spontaneous abortions, stillbirths, elective terminations, minor congenital anomalies, and any serious adverse pregnancy outcomes among pregnancies exposed to Cymbalta and their live births during the first year of life | maximum of 22 months
To examine any potential impact of Cymbalta use while breastfeeding on the infant during the first year of life | maximum of 22 months
To compare the risk of major congenital anomalies among pregnancies exposed to Cymbalta to an appropriate comparator(s) such as the Centers for Disease Control and Prevention (CDC) Metropolitan Atlanta Congenital Defects Program (MACDP) | maximum of 22 months

CONTACTS AND LOCATIONS:
Overall Officials: INC Research, LLC, Study Director — Syneos Health
Locations (1):
- The Cymbalta Pregnancy Registry Call Center, Wilmington, North Carolina, United States